CLINICAL TRIAL: NCT02667938
Title: A Multicenter, Randomized, Double-blind, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of HCP1303 Capsules
Brief Title: A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of HCP1303 Capsules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-TASU-301
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1 (Experimental): HCP1303 capsule 5/0.2mg + HCP1303 capsule 5/0.4mg placebo+ HGP1201 placebo
  Interventions: Drug: HCP1303 capsule 5/0.2mg; Drug: HCP1303 capsule 5/0.4mg placebo; Drug: HGP1201 placebo
- Treatment 2 (Experimental): HCP1303 capsule 5/0.2mg placebo+ HCP1303 capsule 5/0.4mg + HGP1201 placebo
  Interventions: Drug: HCP1303 capsule 5/0.4mg; Drug: HCP1303 capsule 5/0.2mg placebo; Drug: HGP1201 placebo
- Active Comparator (Active Comparator): HCP1303 capsule 5/0.2mg placebo+ HCP1303 capsule 5/0.4mg placebo+ HGP1201
  Interventions: Drug: HGP1201; Drug: HCP1303 capsule 5/0.2mg placebo; Drug: HCP1303 capsule 5/0.4mg placebo

INTERVENTIONS:
Drug: HCP1303 capsule 5/0.2mg
  Arms: Treatment 1
Drug: HCP1303 capsule 5/0.4mg
  Arms: Treatment 2
Drug: HGP1201
  Arms: Active Comparator
Drug: HCP1303 capsule 5/0.2mg placebo
  Arms: Active Comparator; Treatment 2
Drug: HCP1303 capsule 5/0.4mg placebo
  Arms: Active Comparator; Treatment 1
Drug: HGP1201 placebo
  Arms: Treatment 1; Treatment 2

SUMMARY:
The main objective of this study is to evaluate efficacy and safety of HCP1301 capsule in patients with Benign Prostatic Hyperplasia and Erectile Dysfunction

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, phase 3 clinical trial to evaluate the efficacy and safety of HCP1303 capsule

ELIGIBILITY:
Inclusion Criteria:

* At Visit 1

  1. ≥50 age
  2. BPH(Benign Prostatic Hyperplasia) + Total IPSS(International Prostate Symptom Score) ≥ 13
  3. Abnormal Erectile function ≥ at least 3months based on screening date
* At Visit 2 1. Total IPSS ≥ 13

Exclusion Criteria:

1. History of hypersensitivity to Tamsulosin or Tadalafil
2. History of allergy for Sulfonamide
3. PSA (Prostate Specific Antigen) ≥4ng/mL

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change of Total IPSS (International Prostate Symptom Score) | baseline and 12 weeks

SECONDARY OUTCOMES:
Change of Total IPSS | baseline and 4weeks, 8sweeks

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kim, M.D.,Ph.D., Principal Investigator — Catholic University of Seoul St.Mary's Hospital

IPD SHARING:
Plan to Share IPD: No